CLINICAL TRIAL: NCT07293130
Title: Protocol for a Pragmatic, Randomized Controlled, Parallel-group Superiority Trial Comparing the Effectiveness of Mechanical Diagnosis and Therapy Versus Generalized Exercise for Reducing Pain in Surgeons With Chronic Spinal Pain and a Directional Preference
Brief Title: Protocol for a Randomized Controlled Trial Comparing the Effectiveness of Mechanical Diagnosis and Therapy Versus Generalized Exercise for Reducing Pain in Surgeons With Chronic Spinal Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claus Kjærgaard (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Claus Kjærgaard, Principal Investigator; PhD Student, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240046
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spinal Pain
Keywords: spinal pain; chronic pain; musculoskeletal pain; occupational health; surgeons; rehabilitation; exercise
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Masking Description: Outcome assessors and statisticians will remain blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Diagnosis and Therapy (MDT) (Experimental): Individualized exercise-based rehabilitation delivered according to the Mechanical Diagnosis and Therapy (McKenzie) system. Direction-specific exercises are prescribed following a standardized MDT assessment to identify directional preference; progression follows the MDT stages (Reduction → Maintenance of Reduction → Recovery of Function → Prophylaxis). Participants receive education and ergonomic guidance relevant to surgical work. Up to 6 clinic visits over 26 weeks (initial ≈60 minutes; subsequent ≈30 minutes); home exercises prescribed and progressed.
  Interventions: Behavioral: Mechanical Diagnosis and Therapy (MDT)
- Generalized Exercise (Active Comparator): Non-direction-specific, guideline-based exercise rehabilitation focusing on strengthening, flexibility, and endurance to address chronic spinal pain. Program is individualized to symptoms and capacity but does not target directional preference. Participants receive education and ergonomic guidance. Up to 6 clinic visits over 26 weeks (initial ≈60 minutes; subsequent ≈30 minutes); home exercises prescribed and progressed.
  Interventions: Behavioral: Generalized Exercise

INTERVENTIONS:
Behavioral: Mechanical Diagnosis and Therapy (MDT) — Standardized MDT assessment to determine directional preference, followed by direction-specific repeated movements and/or sustained positions. Treatment is progressed across MDT stages (Reduction, Maintenance of Reduction, Recovery of Function, Prophylaxis). Includes brief education, self-management strategies, and occupational ergonomic advice. Delivered by physiotherapists credentialed in MDT (minimum 3 years' experience). Dose/Duration: Up to 6 sessions over 26 weeks (1 × ~60 min intake; ≤5 × ~30 min follow-ups) plus daily home exercises.
  Arms: Mechanical Diagnosis and Therapy (MDT)
Behavioral: Generalized Exercise — Non-direction-specific exercise program comprising progressive strengthening, stretching, and endurance training (e.g., bodyweight, resistance bands, light free weights), paced and progressed according to symptoms and capacity. Includes brief education, self-management strategies, and occupational ergonomic advice. Delivered by physiotherapists experienced in chronic musculoskeletal pain (minimum 3 years' experience). Dose/Duration: Up to 6 sessions over 26 weeks (1 × ~60 min intake; ≤5 × ~30 min follow-ups) plus daily home exercises.
  Arms: Generalized Exercise

SUMMARY:
Surgeons often experience long-lasting spinal pain because of the physical demands of their work, such as long hours in fixed postures and repetitive movements. Chronic pain in the back, neck, or thoracic spine is common, and it can affect health, career longevity, and surgical performance. There is an urgent need for safe and effective non-invasive treatments. Exercise is widely recommended, but it is not clear which type of exercise works best for surgeons with chronic spinal pain.

This clinical trial will compare two exercise approaches: Mechanical Diagnosis and Therapy (MDT), also known as the McKenzie Method, and a structured program of generalized exercise. MDT uses a detailed assessment to identify the direction of movement that reduces pain (called "directional preference") and then prescribes targeted exercises. Generalized exercise includes strengthening, stretching, and endurance training that are not tailored to directional preference. Both treatments are delivered by experienced physiotherapists in real-world outpatient settings.

The main question this study will answer is:

Does MDT reduce pain intensity more than generalized exercise after 12 weeks?

The study will also look at whether these treatments improve daily function, quality of life, work ability, and psychological factors such as fear of movement and pain coping.

Participants will be surgeons aged 25 to 70 years who have had spinal pain for more than three months and who demonstrate a directional preference during assessment. After screening and informed consent, participants will be randomly assigned, like flipping a coin, to one of the two treatment groups.

Participants will:

Attend up to six physiotherapy sessions over 26 weeks.

Receive education, ergonomic advice, and home exercise instructions.

Complete online questionnaires on pain, function, work ability, and quality of life at baseline, 4 weeks, 12 weeks, and 26 weeks.

The primary outcome is the average spinal pain intensity reported on a 0-10 scale after 12 weeks. Secondary outcomes include self-reported function, health-related quality of life, fear of movement, pain catastrophizing, self-efficacy, exercise adherence, therapeutic alliance, impression of change, medication use, and any adverse events.

The study will recruit 60 surgeons in Denmark and follow them for 26 weeks. The trial is designed to be pragmatic, meaning it is carried out under conditions similar to everyday clinical practice, so the results can be applied in real-world settings.

This is the first trial, to our knowledge, that directly compares MDT with a credible, guideline-recommended generalized exercise program in a homogeneous group of surgeons with chronic spinal pain and a directional preference. The findings will provide new evidence on the effectiveness of personalized exercise strategies versus generalized exercise in this high-risk occupational group. If MDT proves to be more effective, it could help improve surgeons' health and their ability to work, while reducing reliance on more invasive or costly interventions.

DETAILED DESCRIPTION:
Chronic spinal pain is highly prevalent among surgeons, who are exposed to long operating hours, static postures, and ergonomic strain. This condition threatens not only personal health but also professional capacity and career longevity. Current evidence supports exercise therapy as a first-line intervention for chronic spinal pain, yet no specific form of exercise has consistently demonstrated superiority. The Mechanical Diagnosis and Therapy (MDT) system, also known as the McKenzie Method, offers a classification-based approach to exercise prescription that may enhance effectiveness in selected patient subgroups. MDT emphasizes the concept of "directional preference," whereby repeated movements in a specific direction lead to rapid and sustained improvements in pain and function. Despite encouraging results from systematic reviews, the evidence base for MDT remains limited, particularly outside the low back pain population, and high-quality randomized controlled trials are needed.

This trial is a pragmatic, randomized, controlled, parallel-group superiority study designed to compare MDT with generalized exercise in surgeons with chronic spinal pain who demonstrate a directional preference. The pragmatic design was chosen to maximize external validity and reflect real-world clinical practice. The study targets a high-risk occupational group and aims to address existing gaps in the literature, including heterogeneous populations, varied therapist training, and limited follow-up durations in prior studies.

Trial design and setting The trial will recruit 60 surgeons in Denmark, working across different surgical specialties. Eligible participants must have experienced spinal pain (cervical, thoracic, or lumbar) for more than three months and demonstrate a directional preference during a standardized physiotherapy assessment. Participants will be randomized 1:1 to MDT or generalized exercise, stratified by sex, with allocation concealed via REDCap. Outcome assessors and statisticians will remain blinded to treatment allocation. The intervention will be delivered in outpatient physiotherapy clinics across Denmark.

Interventions

MDT group: Participants will undergo a structured MDT assessment and receive individualized, direction-specific exercise prescriptions, education, and ergonomic advice. Treatment will follow the four MDT stages (Reduction, Maintenance, Recovery of Function, and Prophylaxis). All therapists will be credentialed in MDT and experienced in clinical application.

Generalized exercise group: Participants will receive non-direction-specific rehabilitation including strengthening, stretching, and endurance training based on current clinical guidelines. Programs will be tailored to participant needs and preferences but will not target directional preference.

Both groups will receive up to six physiotherapy sessions over 26 weeks, including one initial 60-minute session and subsequent 30-minute follow-ups. Written instructions and ergonomic guidance will be provided, and adherence will be reinforced at each visit.

Study objectives The primary objective is to compare the effectiveness of MDT versus generalized exercise in reducing average spinal pain intensity at 12 weeks, measured by the Numeric Pain Rating Scale (NPRS). Secondary objectives include comparing effects on functional limitations, health-related quality of life, psychological variables (fear-avoidance, catastrophizing, self-efficacy), therapeutic alliance, and exercise adherence, as well as recording analgesic use and adverse events.

Rationale for comparator Generalized exercise was chosen as the comparator because it is guideline-recommended, widely used in physiotherapy practice, and represents an ethically justified and clinically credible standard of care. This ensures that the trial tests MDT against a real-world comparator of high external validity.

Sample size and analysis Based on a minimal clinically important difference of 1.5 points on the NPRS and a standard deviation of 2.0, 56 participants (28 per arm) are required to provide 80% power with a two-sided alpha of 0.05. Allowing for 10% attrition, the total recruitment target is 60. Data will be analyzed using linear mixed models with group, time, and their interaction as fixed effects, adjusted for baseline pain. Analyses will follow the intention-to-treat principle, with sensitivity analyses conducted to address missing data.

Blinding Due to the nature of the interventions, participants and treating physiotherapists cannot be blinded. However, outcome collection is self-reported via secure online systems, and statisticians will remain blinded throughout analysis.

Safety and monitoring Both interventions are considered minimal risk, as they are non-invasive physiotherapy treatments delivered by experienced clinicians. Adverse events will be monitored and categorized as serious or non-serious. There is no independent data monitoring committee due to the low-risk nature of the trial, and no interim analyses are planned. Treatments may be modified or discontinued in case of adverse effects, participant request, or medical contraindications.

Significance This is the first randomized controlled trial to compare MDT with a structured, credible generalized exercise program in a homogenous occupational group of surgeons with chronic spinal pain and directional preference. By focusing on a subgroup likely to respond to MDT, standardizing therapist expertise, and implementing a pragmatic multicenter design, this trial aims to provide robust evidence with direct clinical and occupational relevance. If MDT demonstrates superior effectiveness, the findings could inform future guidelines and contribute to improved non-invasive management strategies for spinal pain in high-demand professions.

ELIGIBILITY:
Inclusion Criteria:

Age 25-70 years. Currently working as a resident, fellow, or attending surgeon. Chronic spinal pain (low back, thoracic, or neck) lasting >3 months. Demonstrated directional preference on standardized clinical examination. Sufficient proficiency in Danish to complete trial questionnaires. Willing and able to attend treatment sessions at designated physiotherapy clinics.

Provide written, informed consent.

Exclusion Criteria:

Serious spinal pathology (e.g., fracture, malignancy, infection, inflammatory disease).

Cauda equina syndrome. Significant neurological deficits requiring urgent medical attention. Any diagnosed medical condition preventing safe physical activity. Sick leave >6 months at baseline. Pregnancy or having given birth within the past 3 months. Scheduled for major surgery within the next 3 months. Current participation in structured physiotherapy or spinal interventions outside the trial protocol.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Spinal pain intensity | The primary analysis metric is the change score (12-week NPRS minus baseline NPRS)
  Participant-reported average spinal pain over the past 7 days using the 11-point Numeric Pain Rating Scale (0 = no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Patient-Specific Functional Scale | Baseline, 4 weeks, 12 weeks, 26 weeks
  Self-reported functional limitations; total PSFS score analyzed as change from baseline by group mean
Short Form-12 | Baseline, 4 weeks, 12 weeks, 26 weeks
  Health-related quality of life measured with the SF-12 questionnaire. Scores will be analyzed as change from baseline by group mean. Both Physical Component Summary (PCS) and Mental Component Summary (MCS) scores will be analyzed.
Fear-Avoidance Beliefs Questionnaire | Baseline, 4 weeks, 12 weeks, 26 weeks
  Fear of movement/work; total FABQ score analyzed as change from baseline by group mean
Pain Catastrophizing Scale | Baseline, 4 weeks, 12 weeks, 26 weeks
  Pain catastrophizing; total PCS score analyzed as change from baseline by group mean
Pain Self-Efficacy Questionnaire | Baseline, 4 weeks, 12 weeks, 26 weeks
  Pain self-efficacy; total PSEQ score analyzed as change from baseline by group mean
Working Alliance Inventory | 4 weeks, 12 weeks, 26 weeks (no baseline)
  Therapeutic alliance; total WAI score analyzed as change from prior assessment by group mean
Exercise Adherence Rating Scale | 4 weeks, 12 weeks, 26 weeks (no baseline)
  Exercise adherence; total EARS score analyzed as change from prior assessment by group mean
Patient Global Impression of Change | 4 weeks, 12 weeks, 26 weeks (no baseline)
  Global impression of change; PGIC analyzed by group mean at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Claus Kjærgaard, M.Sc. Health Science, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying published results (text, tables, figures, appendices) will be made available beginning 6 months after publication and for up to 5 years. Access will be granted for academic purposes upon reasonable request through a formal application to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data and supporting documents will be available beginning 6 months after publication of trial results and remain available for 5 years.
Access Criteria: Data will be shared with qualified researchers for academic purposes only. Access requires submission of a reasonable request and a formal application to the Principal Investigator. Approved applicants will receive de-identified data and supporting materials through secure data transfer.
URL: https://vbn.aau.dk